CLINICAL TRIAL: NCT06150092
Title: Use of Presepsin for Early Diagnosis of Sepsis in the Emergency Room
Brief Title: Use of Presepsin in the Emergency Department
Acronym: P-SEP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Piccioni Andrea, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 5984
Record Dates: First submitted 2023-11-16; First posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Sepsis
Keywords: suspected sepsis; early diagnosis of sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sepsis is an extremely common systemic condition in the Emergency Room (ER), which is found to be to be one of the leading causes of death among patients accessing the ER.

To date, the diagnosis of sepsis does not rely on any specific markers for infectious conditions, but several methods of assessing the general condition of the patient, namely markers that elevate in a variety of inflammatory conditions (PCR, PCT), indices of tissue hypoxia (serum lactate), and scores based on the haemochromocytometric examination, the markers of function of different organs, and vital parameters expressed by the patient at the time of assessment (SOFA, qSOFA, SIRS, NEWS). These markers, in addition to not be specific for sepsis, have an insufficiently early peak of presentation to readily identify all patients presenting with this condition.

Presepsin, as the N-terminal portion of the soluble component of Cluster of Differentiation 14 (CD14), is elevated almost exclusively in infectious conditions; moreover, its elevation in infectious contexts is extremely early compared with that of markers already in use, allowing early identification of septic patients who to date would be recognized as such only hours after the onset of the septic process. In addition, the determination of this biomarker could make it possible to stratify patients by prognosis, allowing greater attention to be paid to the most severe patients.

It is hypothesized that the Presepsin assay in emergency room will allow to increase the rapidity and specificity of sepsis diagnosis compared with the diagnostic procedure currently used, improving the outcomes of patients accessing the emergency room with symptoms suggestive of sepsis.

The main purpose of the present study is to evaluate the role of serum assay of presepsin in the early diagnosis of sepsis in patients presenting to the emergency department with clinical suspicion of sepsis by comparing the values obtained with traditionally used such as PCR, PCT, and blood culture. The secondary objective is to evaluate presepsin as a prognostic biomarker and useful for mortality risk stratification of the same patients, comparing the values obtained with validated predictor scores of mortality and/or severity (APACHEII, SOFA, qSOFA).

DETAILED DESCRIPTION:
Study design: Prospective observational study without drug or device

Sample definition: 300 consecutive patients will be included in the study who enter the emergency department with symptoms suggestive of sepsis and who meet the criteria for eligibility. The blood sampling required for the presepsin assay will take place concurrently with the blood draws required for routine testing. Assuming that approximately 70 percent of patients will have a confirmed diagnosis of sepsis and assuming an Area Under the Roc Curve (AUC) of 0.80 this number of patients will allow the AUC of presepsin dosing to be estimated with a 95% confidence interval of overall magnitude of 0.10, thus obtaining an estimate interval from 0.75 to 0.85

Duration of the study: The duration of the study will be 18 months from the approval of the this protocol by the Territorial Ethics Committee (TEC). The enrollment phase of the patients will last 12 months, while the next 6 months will be devoted to data extraction, statistical analysis and scientific reporting.

Procedures: Prospectively enrolled patients will be selected by the attending physician at the time of the first visit and, if eligible, will be asked for written informed consent to participation in the study. Patients will be enrolled during emergency evaluation as part of standard care in the EM, and during blood draws as required by clinical practice routine practice a venous blood sample will be taken at the time of the visit. It will be performed serum analysis and presepsin assay obtained, without additional blood draws.

Variables of interest:

* Presepsin: a peripheral blood sample will be collected by blood sampling and its blood concentration will be assayed in the highly automated CoreLab of the Polyclinic A. Gemelli in Rome.
* Serum lactate: if part of the patient's diagnostic therapeutic pathway, it will be dosed directly in the ER through the device "Hemogasanalyzer pO2 ABL90 FLEX" present in the ER.
* History: will be collected by the ER physician who visits the patient
* Scores: will be calculated based on clinical data obtained during the stay in the ER
* Serum creatinine, PCR, PCT, CBC examination, blood culture and urinocultures: Collection of biological material will be carried out in the emergency room of the A. Gemelli University Polyclinic in Rome, IRCCS; laboratory evaluation and storage of biological material for molecular analysis for the current study will be carried out at the highly automated CoreLab of University Polyclinic A. Gemelli of Rome, IRCCS
* Length of visit to the ER.
* Complications during the stay in the ER and possible admission to intensive care unit or death from any cause

Amendments to the protocol: Any amendments to the protocol will be promptly communicated to the Ethics Committee by the investigators. This will configure the request for additional informed consent, which will be submitted to all patients included in the study.

Error:

* Incorrect association between blood sample and patient;
* insufficient sample for laboratory evaluation
* errors in the laboratory report
* errors in data storage

These possible errors will be minimized by the establishment of specific procedures

related to the study.

Confounding factors: Presepsin values increase:

* In cases of renal failure, but recent studies allow its value to be framed in light of renal function.
* In pediatric age, but our study includes only adult patients.
* In noninfected burn cases, which are not included in the study, and which will be identified through a thorough history and objective examination.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years;
* Patients presenting to the emergency department with suspected clinical sepsis
* Patients who submit at the time of the visit will have a venous blood sample taken.
* Signature of written informed consent to participate to the study and the processing of personal data.

Exclusion Criteria:

* Age <18 years;
* Pregnant women
* Refusal to sign written informed consent to participation in the study and the processing of personal data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients entering the emergency department with symptoms suggestive of sepsis will be included in the study if they are of age, not pregnant who meet the predetermined inclusion criteria. The blood draw required for the presepsin assay will occur at the same time as the blood draws required for routine testing, according to intrahospital guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-10-10 (Estimated); Study Completion 2025-04-10 (Estimated)

PRIMARY OUTCOMES:
Role of serum dosage of presepsin | 3 days
  To evaluate the role of serum dosage of presepsin in the early diagnosis of sepsis in patients presenting to the emergency department with clinical suspicion of sepsis by comparing the values obtained with biomarkers traditionally used

SECONDARY OUTCOMES:
Presepsin as a biomarker prognosticator and predictor of mortality | 30 days
  To evaluate presepsin as a prognostic biomarker and useful for mortality risk stratification of the same patients, comparing the values obtained with validated predictor scores for mortality and/or severity

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario "A. Gemelli" IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No